CLINICAL TRIAL: NCT01682616
Title: A Phase 1b Study Evaluating the Safety and Tolerability of ABT-199 in Combination With Rituximab in Subjects With Relapsed Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M13-365
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2012-06-26; First posted 2012-09-11 (Estimated); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Small Lymphocytic Lymphoma; Chronic Lymphocytic Leukemia
Keywords: Safety; Small Lymphocytic Lymphoma; Chronic Lymphocytic Leukemia; Rituximab; Tolerability; Pharmacokinetics; ABT-199; Cancer; Preliminary; Efficacy; Maximum Tolerated Dose; Venetoclax
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — venetoclax; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Experimental): Chronic Lymphocytic Leukemia (CLL), Small Lymphocytic Lymphoma (SLL)
  Interventions: Drug: ABT-199; Drug: Rituximab

INTERVENTIONS:
Drug: ABT-199 — ABT-199 is taken continuously once daily. This is a dose escalation study, therefore the dose of ABT-199 will change throughout the study.
  Other Names: venetoclax
Drug: Rituximab — Rituximab will be given by intravenous infusion on day 1 of Months 1, 2, 3, 4, 5, and 6. May be reinitiated for an additional 6 months.

SUMMARY:
This is a Phase 1b, open-label, multicenter study evaluating the safety and tolerability of ABT-199 in combination with rituximab in up to 50 subjects with Relapsed Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma. The primary objectives of this study are to assess the safety profile, to determine the maximum tolerated dose and establish the Recommended Phase Two Dose of ABT-199 when administered in combination with rituximab. The dose escalation portion of the study will include approximately 30 subjects. Once the recommended phase two dose and schedule have been determined, up to 20 additional subjects will be enrolled in an expanded safety portion of the study. Subjects who meet criteria for CR, CRi, or MRD-negative PR during the study may discontinue ABT 199. If disease progression occurs, as defined by iwCLL NCI/WG criteria for tumor response, or MRD progression, subjects may re-initiate ABT-199.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be greater then or equal to 18 years of age.
* Subject must have relapsed Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma.
* Subject has an Eastern Cooperative Oncology Group performance score of less than or equal to 1.
* Subject must have adequate bone marrow independent of growth factor support per local laboratory reference range at Screening.
* Subject must have adequate coagulation, renal, and hepatic function, per laboratory reference range at Screening.

Exclusion Criteria:

* Chronic lymphocytic leukemia or Small Lymphocytic Lymphoma subject has undergone an allogeneic or autologous stem cell transplant.
* Subject has uncontrolled autoimmune hemolytic anemia or thrombocytopenia.
* Subject has tested positive for human immunodeficiency virus.
* Seropositivity for hepatitis B surface antigen or hepatitis C virus antibody or ribonucleic acid.
* History of severe allergic or anaphylactic reactions to rituximab.
* Subject has received a live viral vaccine within 6 months prior to the first dose of study drug.
* Subject has received a monoclonal antibody for anti-neoplastic intent within 8 weeks prior to the first dose of study drug.
* Subject has received any of the following within 14 days prior to the first dose of study drug, or has not recovered to less than grade 2 clinically significant adverse effect(s)/toxicity(s) of the previous therapy:

  * Any anti-cancer therapy including chemotherapy, immunotherapy, or radiotherapy;
  * Investigational therapy, including targeted small molecule agents.
* Subject has a cardiovascular disability status of New York Heart Association Class greater then or equal to 2. Class 2 is defined as cardiac disease in which subjects are comfortable at rest but ordinary physical activity results in fatigue, palpitations, dyspnea or anginal pain.
* Subject has a significant history of renal, neurologic, psychiatric, pulmonary, endocrinologic, metabolic, immunologic, cardiovascular, or hepatic disease that in the opinion of the investigator would adversely affect his/her participating in this study.
* Subject has a history of other active malignancies other than CLL/SLL within the past 2 years prior to study entry, with the exception of:

  * Adequately treated in situ carcinoma of the cervix uteri;
  * Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
  * Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent.
* Subject has malabsorption syndrome or other condition that precludes enteral route of administration.
* Subject exhibits evidence of other clinically significant ongoing or recent condition(s) including, but not limited to:

  * Ongoing systemic infection (viral, bacterial, or fungal);
  * Diagnosis of fever and neutropenia within 1 week prior to study drug administration

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-07-25 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Assess the safety profile, to determine the maximum tolerated dose and Recommended Phase Two Dose of ABT-199 when administered in combination with rituximab (R) in subjects with relapsed chronic lymphocytic leukemia and small lymphocytic lymphoma. | Continuous dosing at designated dose level up to Month 6. At end of combination treatment, ABT-199 monotherapy may continue up to 8 years following the date of the last subject enrolled. If disease progression occurs, subjects may re-initiate ABT-199.
  Protocol-defined events, which are attributed as having a reasonable possibility of being related to the administration of ABT-199 and/or rituximab, or can not be attributed by the investigator to a clearly identifiable cause such as tumor progression, concurrent illness, underlying disease or concomitant medication, will be considered a dose limiting toxicity.

SECONDARY OUTCOMES:
Determination of peak concentration (Cmax) of ABT-199 and/or Rituximab. | PK samples collected up to Month 6 for ABT-199 and Rituximab
  Blood samples for analysis of ABT-199 and rituximab will be collected at designated time points.
Assess the exploratory efficacy of the combination ABT-199 and rituximab. | Tumor Assessments will be performed at: Screening, Day 1 on Months 1, 3, 7, and then every 3 months thereafter up to 8 years following the date of the last subject first dose.
  Tumor response or clinical disease progression (Objective Response Rate)
Determination of trough concentration (Ctrough) of ABT-199 and/or Rituximab | PK samples collected up to Month 6 for ABT-199 and Rituximab
  Blood samples for analysis of ABT-199 and rituximab will be collected at designated time points.
Determination of area under the concentration versus time curve (AUC) of ABT-199 and/or Rituximab | PK samples collected up to Month 6 for ABT-199 and Rituximab
  Blood samples for analysis of ABT-199 and rituximab will be collected at designated time points.
Assess the exploratory efficacy of the combination ABT-199 and rituximab | Tumor Assessments will be performed at: Screening, Day 1 on Months 1, 3, 7, and then every 3 months thereafter up to 8 years following the date of the last subject first dose.
  Tumor response or clinical disease progression for (Overall Survival)
Assess the exploratory efficacy of the combination ABT-199 and rituximab | Tumor Assessments will be performed at: Screening, Day 1 on Months 1, 3, 7, and then every 3 months thereafter up to 8 years following the date of the last subject first dose.
  Tumor response or clinical disease progression for (Progression Free Survival)
Assess the exploratory efficacy of the combination ABT-199 and rituximab | Tumor Assessments will be performed at: Screening, Day 1 on Months 1, 3, 7, and then every 3 months thereafter up to 8 years following the date of the last subject first dose.
  Tumor response or clinical disease progression for (Time to Tumor Progression)
Assess the exploratory efficacy of the combination ABT-199 and rituximab | Tumor Assessments will be performed at: Screening, Day 1 on Months 1, 3, 7, and then every 3 months thereafter up to 8 years following the date of the last subject first dose.
  Tumor response or clinical disease progression for (Duration Of Response)

OTHER OUTCOMES:
Assess the exploratory pharmacodynamics and pharmacogenetics of the combination of ABT-199 and rituximab. | MRD Assessments will be performed at following timepoints: At least 2 months after CR/CRi criteria for tumor response first met, every 12 weeks thereafter until MRD negativity is achieved, and as needed.
  Minimal residual disease (MRD) will be assessed in the peripheral blood and bone marrow (BM) either by flow cytometry or real-time PCR.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (6):
- United States (4):
  - Moores Cancer Center at UC San Diego /ID# 70398, La Jolla, California
  - Northwestern University Feinberg School of Medicine /ID# 71593, Chicago, Illinois
  - North Shore University Hospital /ID# 71813, New Hyde Park, New York
  - Duke Cancer Center /ID# 71393, Durham, North Carolina
- Australia (2):
  - Peter MacCallum Cancer Ctr /ID# 70394, Melbourne, Victoria
  - The Royal Melbourne Hospital /ID# 70393, Parkville, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Badawi M, Chen X, Marroum P, Suleiman AA, Mensing S, Koenigsdorfer A, Schiele JT, Palenski T, Samineni D, Hoffman D, Menon R, Salem AH. Bioavailability Evaluation of Venetoclax Lower-Strength Tablets and Oral Powder Formulations to Establish Interchangeability with the 100 mg Tablet. Clin Drug Investig. 2022 Aug;42(8):657-668. doi: 10.1007/s40261-022-01172-4. Epub 2022 Jul 13. PMID 35829925
- [Derived] Roberts AW, Ma S, Kipps TJ, Coutre SE, Davids MS, Eichhorst B, Hallek M, Byrd JC, Humphrey K, Zhou L, Chyla B, Nielsen J, Potluri J, Kim SY, Verdugo M, Stilgenbauer S, Wierda WG, Seymour JF. Efficacy of venetoclax in relapsed chronic lymphocytic leukemia is influenced by disease and response variables. Blood. 2019 Jul 11;134(2):111-122. doi: 10.1182/blood.2018882555. Epub 2019 Apr 25. PMID 31023700
- [Derived] Seymour JF, Ma S, Brander DM, Choi MY, Barrientos J, Davids MS, Anderson MA, Beaven AW, Rosen ST, Tam CS, Prine B, Agarwal SK, Munasinghe W, Zhu M, Lash LL, Desai M, Cerri E, Verdugo M, Kim SY, Humerickhouse RA, Gordon GB, Kipps TJ, Roberts AW. Venetoclax plus rituximab in relapsed or refractory chronic lymphocytic leukaemia: a phase 1b study. Lancet Oncol. 2017 Feb;18(2):230-240. doi: 10.1016/S1470-2045(17)30012-8. Epub 2017 Jan 13. PMID 28089635
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=M13-365#additional-resources-section